CLINICAL TRIAL: NCT01510600
Title: Alternative Lengthening of Telomeres (ALT) in Neuroblastoma
Brief Title: Studying Biomarkers in Samples From Patients With High-Risk Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL12B5; COG-ANBL12B5 (Other: Children's Oncology Group); CDR0000722061 (Other: Clinical Trials.gov); ANBL12B5 (Other: Children's Oncology Group); NCI-2012-00109 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-01-11; First posted 2012-01-16 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Neuroblastoma
Keywords: stage 4S neuroblastoma; localized resectable neuroblastoma; localized unresectable neuroblastoma; recurrent neuroblastoma; regional neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in samples from patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish telomere length measurement by quantitative polymerase chain reaction (qPCR) as an alternative lengthening of telomeres (ALT) detection method in neuroblastoma (NB).
* To determine the frequency of ALT in high-risk NB and the characteristics of ALT+ NB.
* To establish C-circle (extra-chromosomal telomeric DNA circles) level as a marker of ALT activity in NB.
* To evaluate the prognostic significance of ALT in NB.
* To evaluate the utility of the C-circle assay for the detection of circulating tumor DNA in NB patients with an ALT+ tumor.

OUTLINE: Archived tumor tissue and serum samples are analyzed for telomere length measurement, frequency, and C-circle levels by PCR. Results are then compared with patients' age at diagnosis and outcomes including survival data (event-free and overall survival).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Snap-frozen neuroblastoma (NB) tumors collected at diagnosis (Objectives 1 to 3)

  * High-risk stage 3 or 4 NB AND MYCN non-amplified, i.e., exclude stage 4 infants who are not high-risk

    * Up to five high-risk (> 18 months, unfavorable histology) stage 3/MYCN non-amplified tumors
  * Patients preferably treated on protocol COG-A3973 or similar protocols with myeloablative therapy
  * At least 3 years of follow-up for those with no event (current evidence suggests that ALT+ NBs often relapse late, i.e., 2 years or longer from diagnosis)
* NB tumor DNA collected at diagnosis (Objectives 2 & 3)

  * High-risk stage 3 or 4 NB as for Objective 1, except for MYCN status
  * Stage 4 tumors are preferred; may include up to seven high-risk stage 3 tumors with similar distribution of MYCN-amplified and non-amplified tumors
* Frozen serum from NB patients (Objective 5; 2nd stage of project)

  * Paired serum obtained at diagnosis from patients with ALT+ or ALT- tumors identified in Objective 2

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with neuroblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity, as well as the optimal cut-off, for telomere length (TL) qPCR as an ALT detection method
Frequency and characteristics of ALT in high-risk NB
C-circle level as a marker of ALT activity in NB
Prognostic value of ALT
C-circle assay utility in detecting tumor DNA in the serum of NB patients with an ALT

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Lau, MD, Principal Investigator — Sydney Children's Hospitals Network